CLINICAL TRIAL: NCT01866202
Title: Study of Circulating and Tumor Biomarkers in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/00105
Record Dates: First submitted 2012-04-04; First posted 2013-05-31 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aims: To evaluate the role of monoclonal antibodies in the detection of cancer specific antigens in blood and tumor tissue, and the potential use of these antibodies for future evaluation for therapy. Also, to evaluate the presence of circulating tumor cells (CTCs) and to study EMT (epithelial-mesenchymal) signature changes during chemotherapy.

Methods: To take 20mls of blood from advanced breast cancer patients before a new course of anti-cancer therapy, and another 20mls of blood 3 weeks after treatment. In addition, Consent will be obtained to cut 10-15 tissue sections from their archival tumor specimens. Whenever possible, the blood taking will be timed such that no additional needle prick will be done specifically for the purpose of the study, by coinciding it with standard blood taking which is required for the patient's treatment.

Importance of proposed research to science or medicine:Detection of tumor specific antigens in the blood may potentially reduce the need for more invasive biopsies for confirmation of diagnosis of cancer or follow-up of cancer in the future. The identification and development of antibodies specific to these tumor antigens or markers may offer future therapeutic options, or as a vehicle to deliver cytotoxic therapy. Identification of CTCs as well as understanding the changes that occur in EMT signature in these circulating tumor cells may serve as a means of potential means of prognostication and modification of therapy in the future.

Potential Benefits and Risks: Potential risks to the patient include that of blood taking (pain, feeling faint, infection). Patients will not benefit directly from the study but the knowledge gained may help the management of future patients.

Cancer biomarkers, such as antigens and circulating tumor cells, may be a potential area to developing new methods of diagnosis and treatment of cancer. Monoclonal antibiotics are now able to be identified and isolated that may specifically target progenitors of breast cancer as well as CTCs. The changes that occur to CTCs during treatment may serve as a means of prognostication, as well as allow for therapeutic modifications. Clinical correlative studies into these areas (MAbs and CTCs) will serve to determine the role of these in clinical application in the future.

ELIGIBILITY:
Inclusion Criteria:

* Advanced breast cancer patients whose cancer have progressed and are due to start a new course of anti-cancer therapy.The patient needs to have had previous breast cancer surgery at NUH (lumpectomy or mastectomy) or a diagnostic core biopsy for breast cancer, and consent to allow for blood taking and access to archival tissue.

Exclusion Criteria:

* No available archival tumor specimen at NUH.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with Breast Cancer at National University Hospital (Singapore)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Detection of cancer specific antigens in blood and tumor tissue | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Choo AB, Tan HL, Ang SN, Fong WJ, Chin A, Lo J, Zheng L, Hentze H, Philp RJ, Oh SK, Yap M. Selection against undifferentiated human embryonic stem cells by a cytotoxic antibody recognizing podocalyxin-like protein-1. Stem Cells. 2008 Jun;26(6):1454-63. doi: 10.1634/stemcells.2007-0576. Epub 2008 Mar 20. PMID 18356574
- [Background] Tan HL, Fong WJ, Lee EH, Yap M, Choo A. mAb 84, a cytotoxic antibody that kills undifferentiated human embryonic stem cells via oncosis. Stem Cells. 2009 Aug;27(8):1792-801. doi: 10.1002/stem.109. PMID 19544435